CLINICAL TRIAL: NCT02941809
Title: Open-labeled Dose-extending Placebos as an Adjunct to Methadone Treatment: A Pilot Study
Brief Title: Harnessing Placebo Effects in Methadone Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Annabelle Belcher, Assistant Professor of Psychiatry, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00070829
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Opioid-use Disorder; Opioid-Related Disorders
Keywords: medications for opioid use disorder; methadone
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open-Label Placebo (OLP) (Experimental): Participants who are randomly assigned to group OLP will receive placebo pills. In Phase 1 of the study (first two weeks), participants in this group are given one pill, to be taken concomitant with the methadone. In Phase 2 (3 weeks up to 3 months), OLP participants continue to take the single (morning, or AM) pill, and are given a second pill in a bottle as a take-home. OLP participants will meet with the study team at five time points: at baseline (entry into treatment), 2 weeks post-baseline, and 1-, 2- and 3-months post-baseline.
  Interventions: Behavioral: Open-Label Placebo (OLP)
- Treatment as Usual (TAU) (No Intervention): Participants assigned to TAU will not be given placebo pills, but all interactions with the study team (5 meetings total) will be matched in frequency and length.

INTERVENTIONS:
Behavioral: Open-Label Placebo (OLP) — We are designating this as a behavioral intervention for two reasons: (1) the placebo pill is physiologically inert and is not classified under FDA regulations; and (2) other studies have demonstrated that the efficacy of the placebo pill is strongly dependent on the participants' anticipation of an effect. We are presenting the pill's efficacy in an open and transparent way to the participants, but using a positive frame. We feel that this qualifies the placebo pill use as a behavioral intervention, in the same general category as exercise or relaxation.
  Arms: Open-Label Placebo (OLP)

SUMMARY:
More than 2 million individuals in the United States have an Opioid Use Disorder (OUD). Methadone maintenance treatment is the gold standard of medication-assisted treatment for OUD, but high-dose methadone is associated with cardiotoxicity and respiratory complications, among other side effects. These adverse effects make enhancing the effectiveness of lower doses of methadone an attractive therapeutic goal. Long recognized for its capacity to enhance treatment outcomes for a wide range of neuropsychiatric disorders including pain, the placebo effect offers an as-yet untested avenue to such an enhancement. This approach is particularly compelling given that individuals with substance use disorder tend to have higher salience attribution, and may thereby be more sensitive to placebo effects. Our study combines two promising clinical methodologies-open-label placebo and conditioning-to investigate whether placebo effects can increase the effective potency of methadone in treatment-seeking OUD patients.

DETAILED DESCRIPTION:
A total of 120 newly-enrolled treatment-seeking OUD patients will be randomly assigned to one of two different groups: either methadone plus daily open-label placebo (OLP; treatment group), or methadone/Treatment as Usual (TAU; control). Participants will meet with study team members five times over the course of three months of treatment with methadone (baseline, 2 weeks, and 1, 2 and 3 months post-baseline). Throughout this study time period, methadone dosages will be adjusted by an addiction clinician blind to patient assignment, per standard clinical methods. The primary outcome is methadone dose at three months. Secondary outcomes include self-report of drug use; 3-month urine toxicology screen results; and treatment retention. Exploratory outcomes include several environmental as well as personality factors associated with OUD and with propensity to demonstrate a placebo effect.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 or over)
* Newly-admitted to the methadone treatment program

Exclusion Criteria:

* Pregnancy
* Transfers- patients who have initiated methadone treatment course at another methadone treatment facility
* Hospital transfers- patients who initiated methadone treatment course in a hospital setting
* Criminal justice referral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Three-month dose of methadone | Three months (90 days)
  Mean dose of methadone at 3 months (90 days) post-baseline (entry into treatment) will be evaluated for each of the two arms.

SECONDARY OUTCOMES:
Treatment Retention | 90 and 180 days post-baseline (entry into treatment)
  Three-month (90-day) and 6-month (180 day) treatment retention as a binomial (yes/no) variable outcome
Total number of days retained in treatment | One year post-baseline (entry into treatment)
  Total number of days retained in methadone treatment, up to 365 days
Mean number of days of self-reported drug use | Baseline (entry into treatment), two-weeks post-baseline, and 1-, 2-, and 3-months post-baseline.
  Number of days of self-reported drug use will be obtained at all five study meetings time points (baseline, 2-weeks post-baseline, and 1-, 2-, and 3-months post-baseline) for each of the following substances: opiates, cocaine, benzodiazepines, alcohol, and a single, all-encompassing category of "other drug use".
Urine Testing- Quick-tox Screen | Baseline
  Urine toxicology screening via a point of care Quik-tox screen- panel of 13 drugs to determine the presence (positive/negative) of Cocaine, Opiates, Methamphetamine, Cannabis, Amphetamines, Phencyclidine, Benzodiazepines, Barbiturates, Methadone, Oxycodone, MDMA, Buprenorphine, and Fentanyl.
Craving assessment | Baseline (entry into treatment), two-weeks post-baseline, and 1-, 2-, and 3-months post-baseline.
  An adapted one-item visual-analogue scale to assess drug craving. The scale ranges from 0-100 (0- craving not at all, 50- neutral, 100- Very much).
Objective Opioid Withdrawal Scale (OOWS) | Baseline (entry into treatment), two-weeks post-baseline, and 1-, 2-, and 3-months post-baseline.
  A 13-item clinical assessment of physiological signs of withdrawal conducted by the investigator or a research team member. Scores of 0-1 are given for each item and scores are summed ranging from 0-13.
Subjective Opioid Withdrawal Scale (SOWS) | Baseline (entry into treatment), two-weeks post-baseline, and 1-, 2-, and 3-months post-baseline.
  A 16-item patient self-report instrument to assess common subjective symptoms of craving and withdrawal. Scores of 0-4 are given for each item and total scores are summed ranging from 0-64.
Pittsburgh Sleep Quality Inventory (PSQI) | Baseline (entry into treatment), and 1- and 3-months post-baseline
  A 19-item validated tool to assess sleep quality. The 19 self-rated items are combined to form 7 "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The 7 component scores are then added to added a global score, with a range of 0-21 points.
World Health Organization Quality of Life - Brief (WHOQOL-BREF) Assessment | Baseline (entry into treatment), and 1- and 3-months post-baseline
  The WHOQOL-BREF is a 26-item assessment that produces a quality of life profile with four domain scores and two items that are examined separately. The mean score of items within each domain is used to calculate the domain score, which are then transformed to scale scores. The range of scores is between 15 to 105, with a higher score or number being indicative of a higher quality of life.

OTHER OUTCOMES:
Pain Catastrophising Scale (PCS) | Baseline (entry into treatment), and 1- and 3-months post-baseline
  The PCS is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 0-52. The higher the score, the more catastrophizing thoughts are present. A cutoff of more than 30 points is considered to be clinically relevant.
Compliance | Two-weeks post-baseline, and 1-, 2-, and 3-months post-baseline
  Compliance: a visual-analogue scale rating from 0-100 assessing compliance with instructions to take the placebo pill; higher numbers indicate greater compliance.
Methadone side effects checklist | Two-weeks post-baseline, and 1-, 2-, and 3-months post-baseline
  The Methadone Side Effects Checklist (Longwell B, Kestler RJ & Cox TJ, 1979) assesses severity of of 38 commonly reported methadone treatment-associated side effects. 38 symptoms are rated 1-5 (1="no problem at all"; 5="a very bad problem") for a total possible score of 38-190. Higher total scores indicate higher severity of symptoms.
Cleveland Clinic Constipation Scoring system (CCCS) | Baseline (entry into treatment), two-weeks post-baseline, and 1-, 2-, and 3-months post-baseline
  The CCCS (Agachan, Chen, Pfeifer, Reissman, Wexner, 1996) is an 8-item scale of self-reported severity of symptoms of constipation. A total score is derived, with a possible score of 0-32. Higher total scores indicate higher severity of symptoms.
Adapted credibility/expectancy questionnaire | Baseline (entry into treatment), two-weeks post-baseline, and 1-, 2-, and 3-months post-baseline
  A single-item visual analog scale (0-100) assessment of participant beliefs that the placebo pill would improve symptoms of addiction. Higher scores indicate greater belief/expectation of a beneficial placebo pill effect.
Monetary Choice Questionnaire (MCQ) | Two-weeks post-baseline, and 2-, and 3-months post-baseline
  The MCQ (Kirby & Marakovic, 1996) is a 27-item assessment of delay discounting. For each item, the participant chooses between a smaller, immediate monetary reward and a larger, delayed monetary reward. The protocol is scored by calculating where the respondent's answers place him/her amid reference discounting curves, where placement amid steeper curves indicates higher levels of impulsivity.
Barratt Impulsivity Scale, version 11 (BIS-11) | Two weeks post-baseline
  The BIS-11 (Patton, Stanford, Barratt, 1995) is a 30-item assessment that yields information regarding three facets of trait impulsivity (ie, attentional impulsivity, motor impulsivity and non-planning impulsivity). Participants indicate on a four-point Likert-like scale the extent to which each of 30 items describes their overall behavior. A scoring algorithm (with some items reverse-scored) yields 6 first-order and 3 second-order factors, as well as an overall score (a total possible score of 120). Higher values on each of the factors indicate higher levels of impulsivity.
Exit survey | Three months post-baseline
  A 7-item quantitative and qualitative assessment of how the placebo pill was experienced by participants and their thoughts about their experience participating in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Annabelle M Belcher, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Maryland Methadone Treatment Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belcher AM, Cole TO, Greenblatt AD, Hoag SW, Epstein DH, Wagner M, Billing AS, Massey E, Hamilton KR, Kozak ZK, Welsh CJ, Weintraub E, Wickwire EM, Wish ED, Kaptchuk TJ, Colloca L. Open-label dose-extending placebos for opioid use disorder: a protocol for a randomised controlled clinical trial with methadone treatment. BMJ Open. 2019 Jun 21;9(6):e026604. doi: 10.1136/bmjopen-2018-026604. PMID 31230007
- [Background] Cai NS, Quiroz C, Bonaventura J, Bonifazi A, Cole TO, Purks J, Billing AS, Massey E, Wagner M, Wish ED, Guitart X, Rea W, Lam S, Moreno E, Casado-Anguera V, Greenblatt AD, Jacobson AE, Rice KC, Casado V, Newman AH, Winkelman JW, Michaelides M, Weintraub E, Volkow ND, Belcher AM, Ferre S. Opioid-galanin receptor heteromers mediate the dopaminergic effects of opioids. J Clin Invest. 2019 Mar 26;129(7):2730-2744. doi: 10.1172/JCI126912. PMID 30913037
- [Derived] Belcher AM, Cole TO, Massey E, Billing AS, Wagner M, Wooten W, Epstein DH, Hoag SW, Wickwire EM, Greenblatt AD, Colloca L, Rotrosen J, Magder L, Weintraub E, Wish ED, Kaptchuk TJ. Effectiveness of Conditioned Open-label Placebo With Methadone in Treatment of Opioid Use Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e237099. doi: 10.1001/jamanetworkopen.2023.7099. PMID 37043203